CLINICAL TRIAL: NCT05798169
Title: Impact of Acute Hospitalisation and Resistance Training on Muscle Architecture and Physical Performance in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: University of Copenhagen (Other); Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Lisbeth Rosenbek Minet, Professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARTMAP
Record Dates: First submitted 2022-11-07; First posted 2023-04-04 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Sarcopenia; Functional Decline; Muscle Architecture; Gait Speed; Ultrasound; Physical Performance; Resistance Training; Hospitalisation; Acutely Ill; Older Adults
MeSH Terms: conditions — Sarcopenia | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Group of participants receiving resistance training during hospitalisation
  Interventions: Other: Resistance training
- Control Group (Sham Comparator): Group of participants receiving sham training during hospitalisation
  Interventions: Other: Resistance training

INTERVENTIONS:
Other: Resistance training — Moderate resistance training by a innovative training robot 2 times a day during hospitalisation

SUMMARY:
Sarcopenia characterised by loss of muscle mass, muscle strength and physical performance burdens many older adults since the condition is related to functional decline. Periods of inactivity such as during hospitalisation leads to further functional decline. It has been reported that the loss of muscle mass associated with sarcopenia not only entails a decrease in muscle mass but also changes in muscle architecture. Knowledge on changes in muscle architecture is essential since it is one of the most important determinants on muscle strength and thus physical performance. The main objective of this study is to investigate changes in muscle architecture and physical performance during acute hospitalisation and after discharge in older adults and subsequently the effectiveness of resistance training of the lower limb during acute hospitalisation. If successful, our study could have a great impact on the individual, as well as societal level, due to a better understanding of the factors related to sarcopenia and the prevention of functional decline as a result of hospitalisation.

ELIGIBILITY:
Inclusion Criteria:

* ≥65 years of age
* Able to ambulate before hospitalization (with/without assistance)
* Able to communicate with the research team
* Expected length of stay ≥2 days
* Residing on Funen

Exclusion Criteria:

* Able to ambulate without assistance during current hospitalization
* Known severe dementia
* Positive Confusion and Assessment Method score
* Patients who have received less than 3 resistance training sessions at discharge
* Terminal illness
* Recent major surgery or lower extremity bone fracture in the last 3 months
* Conditions contradicting use of ROBERT(unstable vertebral-, pelvic, or lower extremity fractures
* high intracranial pressure
* pressure ulcers or risk of developing pressure ulcers due to fragile skin
* patients with medical instability)
* Metastases at femur hip
* Deemed not suitable for resistance training sessions with the robot by the healthcare professional.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 274 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline B-mode ultrasonography | Baseline (day of hospitalisation) to day of discharge from hospital (an average of a week).
  Muscle architecture of the m Vastus Lateralis assessed with B-mode ultrasonography.
Change from baseline 4 meter Gait Speed Test | Baseline (Day of hospitalisation) to day of discharge from hospital (an average of a week).
  Physical performance evaluated by the 4m Gait Speed test
Change from baseline B-mode ultrasonography | Change from baseline (day of hospitalisation) to 1-month follow-up and 3-months follow-up
  Muscle architecture of the muscle vastus lateralis assessed with B-mode ultrasonography.
Change from baseline 4 meter Gait Speed Test | Change from baseline (day of hospitalisation) to 1-month follow-up and 3-months follow-up
  Physical performance evaluated by the 4m Gait Speed test

SECONDARY OUTCOMES:
Change from baseline 30s Chair Stand test | Baseline (day of hospitalisation) to day of discharge from hospital (an average of a week)
  Maximal muscle strength of the lower extremities evaluated by the 30s Chair Stand Test or the m30s Chair Stand Test (Modified).
Change from baseline Barthel-Index 100 (Shahs version) | Baseline (day of hospitalisation) to day of discharge from hospital (an average of a week)
  Functional level evaluated by The Barthel-Index 100 (Shahs version)
Change from baseline Bioimpedance | Baseline (day of hospitalisation) to day of discharge from hospital (an average of a week)
  Muscle quantity (kg) on wholebody level evaluated by Bioimpedance
Length of hospital stay | Baseline (day of hospitalisation) to day of discharge from hospital (an average of a week)
  Number of days hospitalised
Mortality | Baseline (day of hospitalization) to 3-months follow-up
  Administrative registers will be used to assess mortality
Unplanned hospitalisation | Day of discharge from hospital to 3-months follow-up
  Patients will be followed through a review of medical records for any unplanned Adminstrative registers will be used to assess any unplanned hospitalisation during the period of inclusion.
Individual level of physiotherapy | Baseline (day of hospitalisation) to 3-months follow-up
  Adminstrative registers and municipalities health records will be used to assess the individual level of physiotherapy (minutes of consultation) in the period of inclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Kristian B Buhl, MD, Study Director — Department of Geriatric, Odense University Hospital
Locations (1):
- Geriatric Deparment OUH Svendborg Hospital, Svendborg, FYN, Denmark

IPD SHARING:
Plan to Share IPD: No
No plan